CLINICAL TRIAL: NCT06935123
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel-Group Study Evaluating Nutritional Supplementation On Sleep Quality
Brief Title: Impact of Nutritional Supplementation on Sleep Quality
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFCRO-189
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Sleep; Sleep Quality
Keywords: sleep; sleep quality; magnesium
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomised, Double-Blind, Placebo-Controlled, Parallel
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sleep Supplement 1 (Active Comparator): Participants served Sleep Supplement 1
  Interventions: Dietary Supplement: Sleep Supplements
- Sleep Supplement 2 (Active Comparator): Participants served Sleep Supplement 2
  Interventions: Dietary Supplement: Sleep Supplements
- Sleep Supplement 3 (Active Comparator): Participants served Sleep Supplement 3
  Interventions: Dietary Supplement: Sleep Supplements
- Sleep Supplement 4 (Active Comparator): Participants served Sleep Supplement 4
  Interventions: Dietary Supplement: Sleep Supplements
- Placebo (Placebo Comparator): Participants served placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sleep Supplements — Sleep supplements
  Arms: Sleep Supplement 1; Sleep Supplement 2; Sleep Supplement 3; Sleep Supplement 4
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 5-arm parallel-group study to evaluate the effects of 4 nutritional supplements on sleep over a 12 week period in healthy U.S. adults.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 18-65 years of age (inclusive).
3. Insomnia severity Index score ≤14.
4. PROMIS Sleep Disturbance Questionnaire raw score ≥23
5. Be willing to maintain stable dietary habits and physical activity levels throughout the study period.
6. Willing to consume the study product daily for the duration of the study.

Exclusion Criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception as determined by the investigator.
3. Has a history of drug and/or alcohol abuse.
4. Hypersensitive to the contents of the study product.
5. Participants with work schedules that result in irregular sleep patterns/ or have night-shift employment.
6. High caffeine intake, >400mg/day.
7. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history. Excluded health conditions include:

   1. Diagnosed Sleep disorders
   2. Major psychiatric diagnosis (e.g., bipolar), as diagnosed by a healthcare professional, including major depressive disorder (e.g., clinical depression)
   3. Immunocompromised health conditions
8. Currently or recently (in the past 4 weeks) taking a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

   1. Prescribed sleep medications
   2. Prescribed Medications which impact sleep, including but not limited to sedative hypnotics, anxiolytics, and antidepressants.
9. Current or recent (in the past 4 weeks) use of prohibited nutritional and non-nutritional supplements with known or possible sleep effects (e.g. valerian, multivitamins, melatonin)
10. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
11. Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-04-11 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance 8A | 0, 4, 8, and 12 weeks
  Perceived sleep quality

SECONDARY OUTCOMES:
PROMIS Sleep Related Impairment 8A | 0, 4, 8, and 12 weeks
  Perceived functional impairments during wakefulness associated with sleep problems or impaired alertness.
Insomnia Severity Index (ISI) | 0, 4, 8, and 12 weeks
  Severity of sleep difficulties and satisfaction with sleep
Depression, Anxiety, and Stress Scale - 21 Items (DASS-21) | 0, 4, 8, and 12 weeks
  Severity of general psychological distress and symptoms related to depression, anxiety, and stress
Bristol Stool Scale (BSS) | 0, 4, 8, and 12 weeks
  Stool frequency and consistency

OTHER OUTCOMES:
Safety Objectives | 0, 4, 8, and 12 weeks
  Occurrence of any Adverse Events (AEs/SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials Inc., 142 E. Ontario, Suite 1200, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No